CLINICAL TRIAL: NCT05213676
Title: Inhaled Nitric Oxide (iNO) for Congenital Diaphragmatic Hernia (CDH) - The "NoNO Trial" - a Multi-center, De-implementation, Stepped-wedge, Cluster-randomized Trial Within an Established Collaborative
Brief Title: De-implementing Inhaled Nitric Oxide for Congenital Diaphragmatic Hernia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: University of Tennessee & LeBonheur Children's Hospital (UT-LBCH) (Unknown); University of California-Irvine & Children's Hospital of Orange County (UC-CHOC) (Unknown); Medical University of South Carolina Children's Health (MUSC) (Unknown); University of Michigan & CS Mott Children's Hospital (UM-CSMott) (Unknown); Randall Children's Hospital-Portland (RCH) (Unknown); Stanford University & Lucile Packard Children's Hospital (Stanford-LPCH) (Unknown); University of California, San Diego & Rady Children's Hospital (UCSD-Rady) (Unknown); Harvard University & Boston Children's Hospital (Harvard-BCH) (Unknown); Indiana University & Riley Children's Hospital (IU-RiCH) (Unknown); University of Louisville & Norton Children's Hospital (UL-NCH) (Unknown); University of Utah & Primary Children's Hospital (Utah-PCH) (Unknown); University of Washington & Seattle Children's Hospital (UW-SCH) (Unknown); University of Alabama & Children's Hospital of Alabama (UAB-CoA) (Unknown); University of Arkansas & Arkansas Children's Hospital (UA-ACH) (Unknown); Vanderbilt University & Vanderbilt University Medical Center (VUMC) (Unknown); University of Southern California & Children's Hospital Los Angeles (USC-CHLA) (Unknown); Emory University & Children's Healthcare of Atlanta (CHOA) (Unknown); University of Colorado & Children's Hospital of Colorado (CU-CHC) (Unknown)
Responsible Party: Principal Investigator, Matthew T Harting, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-21-0603
Record Dates: First submitted 2022-01-27; First posted 2022-01-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Congenital Diaphragmatic Hernia
Keywords: CDH; Inhaled Nitric Oxide; Pulmonary Hypertension
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital; Hypertension, Pulmonary | interventions — Inosine

STUDY DESIGN:
Intervention Model Description: In this multi-center study, centers will use iNO per their usual protocol, and centers will then crossover to iNO de-implementation (that is, at the time of crossover, centers will stop using iNO in the initial resuscitation period). A stepped-wedge crossover study design will be used, and the timing of crossover will be cluster randomized at the level of the center.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inhaled Nitric Oxide (iNO) use (Active Comparator): The center will use iNO per their usual protocol in the initial resuscitation period (defined as birth through stabilization and CDH repair). No center will alter any component of their standard clinical practice guideline or protocol governing CDH care.
  Interventions: Drug: Inhaled Nitric Oxide (iNO) use
- De-implementation of Inhaled Nitric Oxide (iNO) use (Active Comparator): The center will stop using iNO in the initial resuscitation period (defined as birth through stabilization and CDH repair).
  Interventions: Other: De-implementation of Inhaled Nitric Oxide (iNO) use

INTERVENTIONS:
Drug: Inhaled Nitric Oxide (iNO) use — The center will use iNO per their usual protocol in the initial resuscitation period (defined as birth through stabilization and CDH repair). No center will alter any component of their standard clinical practice guideline or protocol governing CDH care.
  Arms: Inhaled Nitric Oxide (iNO) use
Other: De-implementation of Inhaled Nitric Oxide (iNO) use — The center will stop using iNO in the initial resuscitation period (defined as birth through stabilization and CDH repair).
  Arms: De-implementation of Inhaled Nitric Oxide (iNO) use

SUMMARY:
The purpose of this study is to determine if de-implementation of inhaled nitric oxide (iNO) in the post-natal resuscitation/stabilization phase affects the composite outcome of extracorporeal life support (ECLS) use and/or mortality, as well as ECLS use, mortality, and/or oxygenation in congenital diaphragmatic hernia (CDH) newborns and to establish the cost-effectiveness of de-implementing iNO as a therapy in the postnatal resuscitation/stabilization phase of CDH management, which will be assessed as the incremental health system costs (savings) per prevented ECLS use and/or death.

DETAILED DESCRIPTION:
In this multi-center study, centers will use iNO per their usual protocol, and centers will then crossover to iNO de-implementation (that is, at the time of crossover, centers will stop using iNO in the initial resuscitation period). A stepped-wedge crossover study design will be used, and the timing of crossover will be cluster randomized at the level of the center.

ELIGIBILITY:
Inclusion Criteria:

* Postnatal, live born neonates with CDH

  a. Presence of associated or additional anomalies is acceptable for inclusion
* Bochdalek hernia location (right or left)
* Diagnosed prior to 1 month of life
* Born within or transferred to (within 1 week of life) a CDHSG member center participating in the trial

Exclusion Criteria:

* CDH diagnosis after 1 month of age
* Morgagni diaphragmatic hernia (central / anterior-medial diaphragmatic defect location)
* Transferred to a CDH Study Group (CDHSG) member center after 1 week of life
* Patients without potential access to iNO

Ages: 0 Months to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2030-10-31 (Estimated); Study Completion 2031-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who require Extracorporeal Life Support (ECLS) and/or who die prior to discharge | from birth through hospital discharge (up to 12 months from birth)
  The primary outcome is the composite outcome of ECLS use and/or mortality.

SECONDARY OUTCOMES:
Number of participants who require Extracorporeal Life Support (ECLS) prior to discharge | from birth through hospital discharge (up to 12 months from birth)
Number of participants who die prior to discharge | from birth through hospital discharge (up to 12 months from birth)
Change in oxygenation | 1 hour after initiation of iNO use
  For the iNO de-implementation arm, participants will be assessed 1 hour after the time when iNO would have been initiated, per the protocol of the center.
Change in oxygenation | 6 hours after initiation of iNO use
  For the iNO de-implementation arm, participants will be assessed 6 hours after the time when iNO would have been initiated, per the protocol of the center.
Total cost of initial inpatient care from birth through hospital discharge, per center | from birth through hospital discharge (up to 12 months from birth)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Harting, MD, MS, FACS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (19):
- United States (19):
  - University of Alabama & Children's Hospital of Alabama (UAB-CoA), Birmingham, Alabama
  - University of Arkansas & Arkansas Children's Hospital (UA-ACH), Little Rock, Arkansas
  - University of California-Irvine & Children's Hospital of Orange County (UC-CHOC), Irvine, California
  - University of Southern California & Children's Hospital Los Angeles (USC-CHLA), Los Angeles, California
  - Stanford University & Lucile Packard Children's Hospital (Stanford-LPCH), Palo Alto, California
  - University of California, San Diego & Rady Children's Hospital (UCSD-Rady), San Diego, California
  - University of Colorado & Children's Hospital of Colorado (CU-CHC), Aurora, Colorado
  - Emory University & Children's Healthcare of Atlanta (CHOA), Atlanta, Georgia
  - Indiana University & Riley Children's Hospital (IU-RiCH), Indianapolis, Indiana
  - University of Louisville & Norton Children's Hospital (UL-NCH), Louisville, Kentucky
  - Harvard University & Boston Children's Hospital (Harvard-BCH), Boston, Massachusetts
  - University of Michigan & CS Mott Children's Hospital (UM-CSMott), Ann Arbor, Michigan
  - Randall Children's Hospital-Portland (RCH), Portland, Oregon
  - Medical University of South Carolina Children's Health (MUSC), Charleston, South Carolina
  - University of Tennessee & LeBonheur Children's Hospital (UT-LBCH), Memphis, Tennessee
  - Vanderbilt University & Vanderbilt University Medical Center (VUMC), Nashville, Tennessee
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah & Primary Children's Hospital (Utah-PCH), Salt Lake City, Utah
  - University of Washington & Seattle Children's Hospital (UW-SCH), Seattle, Washington

IPD SHARING:
Plan to Share IPD: No